CLINICAL TRIAL: NCT05256147
Title: Effect of Combination Non Steroidal Antiinflammatory Drugs and Narrowband UVB Treatment in Non-Photoadapters
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruiting study population
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9744
Record Dates: First submitted 2017-02-22; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): There is one group in this study and they will receive ibuprofen 400 mg before their narrow band UVB phototherapy session which occurs two to three times weekly. The treatment dose of NBUVB will start off at 150 mJ/cm2 and will be increased 10% as tolerated til the patient reaches 700 mJ/cm2. They will receive ibuprofen before each phototherapy session.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Patient will receive ibuprofen 400 mg before the phototherapy session.

SUMMARY:
Narrow band UVB phototherapy is the mainstay of therapy for vitiligo. However, about 1/3 of patients cannot respond to phototherapy. The objective of this study is to determine if the use of ibuprofen can induce non-photoadapters (patients who cannot tolerate increases in NBUVB past 400 mJ/cm2 after 12 sessions) to convert to photoadapters and tolerate raising NBUVB doses to therapeutic levels

DETAILED DESCRIPTION:
Vitiligo is an acquired disorder of pigmentation. The depigmented regions present as white macules and patches and can occur at any age. The vitiligo patches may be asymptomatic, pruritic or may sunburn. Vitiligo has been shown to significantly impact the quality of life and also has an associated psychological burden. Therefore, treatment of vitiligo is essential. Various treatment modalities such as topical corticosteroids, topical calcineurin inhibitors, systemic steroids, surgery, and phototherapy exist to treat vitiligo. UV based phototherapy includes NBUVB, targeted phototherapy, psoralen and UVA photochemotherapy (1-3).

NBUVB is a proven, effective, and well-accepted treatment as part of the standard of care for vitiligo. NBUVB has a sharp emission peak at 311-313 nm. NBUVB is a relatively safe treatment modality, but can cause phototoxic reactions and tanning. Studies have shown that treatment with NBUVB improves the Vitiligo Area Scoring Index by 42% over a period of 6 months. Approximately half of patients should expect 50% repigmentation by 6 months of 2-3x per week phototherapy (4-6). However, a portion of patients are slow responders requiring up to 72 treatments before notable repigmentation has been achieved.

To complicate matters further, about 1/3 of the patients with vitiligo do not photoadapt, meaning the patient does not exhibit a diminished erythema (redness) to equivalent doses of NBUVB upon future irradiations (7). Photoadaption is the principle behind needing to increase the NBUVB dose for all phototherapy regimens (atopic dermatitis, psoriasis, mycosis fungiodes, vitiligo, etc) and why people are able to tolerate longer solar exposure at the end of summer rather than the beginning. It is thought that the non-photoadapters do not respond to NBUVB as their photoadpative capacity may be genetically predetermined (7).

Repigmentation from NBUVB therapy has shown dramatic improvements in quality of life scores (QOL). Tijoe et. al reported 70% improvement in QOL with long term UVB therapy (8). Therefore, identifying adjunctive therapies that can enable non-photoadapters to safely tolerate therapeutic NBUVB doses can significantly raise their QOL. In addition, these therapies can be expanded into the treatment of photoadapters receiving NBUVB to permit higher dose escalations and fewer phototherapy sessions to achieve a therapeutic NBUVB vitiligo dose. This can in-turn potentially decrease health care costs for increased treatments. Also, the patient may experience fewer long-term side effect associated with NBUVB since they may need fewer sessions of NBUVB.

A possible way for non-photoadapters to tolerate NBUVB may be with the use of NSAIDs. Studies performed have shown that the use of NSAIDs showed increased minimal erythema dose by possibly suppressing the immune response by inhibiting cyclooxygenase and prostaglandins (9). Ibuprofen has also shown to decrease inflammation induced by UVB phototherapy (10). Thus, ibuprofen may increase the MED in non-photoadapters.

Therefore, the goal of this study is to see if the use of ibuprofen, an NSAID, will allow for nonphotoadpaters to respond to NBUVB treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a diagnosis of vitiligo.
* Patients who are identified as nonphotoadapters (those who cannot increase NBUVB dose past 400 mJ/cm2) will be recruited for the study

Exclusion Criteria:

* Patients with the daily ibuprofen use, history of renal disease, cardiac disease, gastric uler and bleeding disorder will be excluded from the study. Patients with a history of lupus erythematosus and other photosensitivity disorders will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
Vitiligo Area Scoring Index (VASI) | 4 months
  Investigator will assess surface area of vitiligo using VASI

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Dermatology, Detroit, Michigan, United States

REFERENCES:
- [Background] Alikhan A, Felsten LM, Daly M, Petronic-Rosic V. Vitiligo: a comprehensive overview Part I. Introduction, epidemiology, quality of life, diagnosis, differential diagnosis, associations, histopathology, etiology, and work-up. J Am Acad Dermatol. 2011 Sep;65(3):473-491. doi: 10.1016/j.jaad.2010.11.061. PMID 21839315
- [Background] Linthorst Homan MW, Spuls PI, de Korte J, Bos JD, Sprangers MA, van der Veen JP. The burden of vitiligo: patient characteristics associated with quality of life. J Am Acad Dermatol. 2009 Sep;61(3):411-20. doi: 10.1016/j.jaad.2009.03.022. Epub 2009 Jul 3. PMID 19577331
- [Background] Hamzavi IH, Lim HW, Syed ZU. Ultraviolet-based therapy for vitiligo: what's new? Indian J Dermatol Venereol Leprol. 2012 Jan-Feb;78(1):42-8. doi: 10.4103/0378-6323.90945. PMID 22199059
- [Background] Hamzavi I, Jain H, McLean D, Shapiro J, Zeng H, Lui H. Parametric modeling of narrowband UV-B phototherapy for vitiligo using a novel quantitative tool: the Vitiligo Area Scoring Index. Arch Dermatol. 2004 Jun;140(6):677-83. doi: 10.1001/archderm.140.6.677. PMID 15210457
- [Background] Scherschun L, Kim JJ, Lim HW. Narrow-band ultraviolet B is a useful and well-tolerated treatment for vitiligo. J Am Acad Dermatol. 2001 Jun;44(6):999-1003. doi: 10.1067/mjd.2001.114752. PMID 11369913
- [Background] Pacifico A, Leone G. Photo(chemo)therapy for vitiligo. Photodermatol Photoimmunol Photomed. 2011 Oct;27(5):261-77. doi: 10.1111/j.1600-0781.2011.00606.x. PMID 21950634
- [Background] Hexsel CL, Mahmoud BH, Mitchell D, Rivard J, Owen M, Strickland FM, Lim HW, Hamzavi I. A clinical trial and molecular study of photoadaptation in vitiligo. Br J Dermatol. 2009 Mar;160(3):534-9. doi: 10.1111/j.1365-2133.2008.08943.x. Epub 2008 Dec 5. PMID 19067714
- [Background] Edwards EK Jr, Horwitz SN, Frost P. Reduction of the erythema response to ultraviolet light by nonsteroidal antiinflammatory agents. Arch Dermatol Res. 1982;272(3-4):263-7. doi: 10.1007/BF00509055. PMID 7165335
- [Background] Stern RS, Dodson TB. Ibuprofen in the treatment of UV-B-induced inflammation. Arch Dermatol. 1985 Apr;121(4):508-12. PMID 3883908